CLINICAL TRIAL: NCT00555009
Title: Placebo Controlled Trial on the Efficacy of Growth Hormone Replacement Therapy in Patients With Growth Hormone Deficiency After Traumatic Brain Injury.
Brief Title: Treatment Of Adult Growth Hormone Deficiency After Traumatic Brain Injury
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6281289
Record Dates: First submitted 2007-10-24; First posted 2007-11-07 (Estimated); Results first posted 2010-06-02 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2009-03

CONDITIONS: Brain Injuries; Growth Hormone Deficiency
Keywords: traumatic brain Injury, cognitive function
MeSH Terms: conditions — Brain Injuries; Dwarfism, Pituitary; Brain Injuries, Traumatic | interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Genotropin treatment arm (Experimental)
  Interventions: Drug: Genotropin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Genotropin — Subcutaneous injection, starting dose 0.2mg/day for males and 0.3mg/day for female with dose titration at 0.1mg to 0.2 mg increments in accordance to IGF-1 results for a total duration of 36 weeks.
  Arms: Genotropin treatment arm
Drug: Placebo — Subcutaneous injection, with dummy dose titration for a total duration of 36 weeks.
  Arms: Placebo

SUMMARY:
To establish the effects of genotropin replacement on cognitive function in patients with severe growth hormone deficiency after traumatic brain injury.

DETAILED DESCRIPTION:
The study was terminated on 15-Dec-2008 due to an inability to recruit the protocol specified patient population. The study has not been terminated due to any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Have had a previous traumatic brain injury (more than 1 year and less than 20 years) prior to the screening visit.
* Have an Extended Glasgow Outcome Scale (GOS-E) more than or equal to 5.
* Have proven GHD deficiency

Exclusion Criteria:

* Active systemic malignancy or active intracranial tumor. A successfully treated tumor or malignancy is not an exclusion criterion if the patient has not had active disease for 5 years and is not currently receiving maintenance chemotherapy, (except for basal cell skin cancers.
* Receiving treatment with prednisolone in doses above 10 mg/day or treatment with other oral glucocorticosteroids above replacement doses is not permitted throughout the study. Topical and inhaled corticosteroids are permitted.
* History of dementia unrelated to TBI
* History of benign intracranial hypertension

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- France (2):
  - Pfizer Investigational Site, Créteil
  - Pfizer Investigational Site, Paris
- Italy (2):
  - Pfizer Investigational Site, Ferrara
  - Pfizer Investigational Site, Roma
- Pfizer Investigational Site, Rotterdam, Netherlands
- Pfizer Investigational Site, Seville, Sevilla, Spain
- Sweden (2):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Stockholm
- Pfizer Investigational Site, Salford, Manchester, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6281289&StudyName=Treatment%20Of%20Adult%20Growth%20Hormone%20Deficiency%20After%20Traumatic%20Brain%20Injury

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to poor recruitment, the study was terminated early; therefore efficacy analyses were not completed.
Groups:
- Genotropin: Initiated at 0.2 mg/day subcutaneously (SC) in men and 0.3 mg/day SC in women. Dose adapted monthly in 0.1 or 0.2 mg increments until stabilized in upper half of normal range.
- Placebo: Matching placebo injected SC.
Period: Overall Study
Arm/Group | Genotropin | Placebo
Started | 4 | 6
Completed | 2 | 0
Not Completed | 2 | 6
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Terminated by Sponsor | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Genotropin | Placebo | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Customized [Number; unit: participants]
  <18 years | 0 | 0 | 0
  18 - 44 years | 4 | 4 | 8
  45-64 years | 0 | 2 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Cognitive Function (CogState™) Composite Score at Week 36
Description: CogState™: 7 tasks: Detection (Part A); Identification; One back working memory; Monitoring; One card learning; Prediction; Detection (Part B). Detection, Identification, Monitoring score range: 2 (worse) to 5 (best); One back working memory/one card learning score range: 0 (worse) to 1.57 (best); Prediction score range: 0 (worse) to 100 (best). Composite change score=average of cognitive change scores for each task at each postdrug assessment; total possible score: -300 to 300. Change=change from baseline (average of 2 postdose assessments). Positive composite score=improved performance.
Time Frame: Baseline, Week 36
Population: Due to poor recruitment, the study was terminated early; therefore efficacy analyses were not completed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Genotropin | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in CogState™ at Week 12 and 24.
Description: as for outcome 1
Time Frame: Baseline, Week 12 and 24
Population: Due to poor recruitment, the study was terminated early; therefore efficacy analyses were not completed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Genotropin | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in Lean Body Mass and Fat Mass at Week 36
Description: The change from Baseline values for lean body mass and fat mass is calculated as the difference between the parameter values at Visit 36, and the parameter values at Baseline.
Time Frame: Baseline, Week 36
Population: Due to poor recruitment, the study was terminated early; therefore efficacy analyses were not completed.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Genotropin | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in Neurological Outcome as Assessed by Extended Glasgow Outcome Scale (GOS-E) at Week 36
Description: The GOS is widely used for assessing outcome after head injury and non-traumatic acute brain insults and is performed by a physician. The GOS-E uses eight points to assess disability and handicap. The GOS-E focuses on how the injury has affected functioning in major areas of life rather than on the particular deficits and symptoms caused by injury. The overall score ranges from 1-8; 1=Death and 8=Upper Good Recovery
Time Frame: Baseline, Week 36
Population: Due to poor recruitment, the study was terminated early; therefore efficacy analyses were not completed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Genotropin | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Quality of Life Using Short Form (SF)-36 Health Survey at Week 36
Description: A subject administered scale assessing general quality of life. A subject administered score, scale, direction of scale. The SF-36 consists of 36 questions covering the following eight health domains (subscales): Physical Functioning, Bodily Pain, Role Limitations Due to Physical Problems, Role Limitations Due to Emotional Problems, General Health Perceptions, Mental Health, Social Function, Vitality.
Time Frame: Baseline, Week 36
Population: Due to poor recruitment, the study was terminated early; therefore efficacy analyses were not completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Genotropin | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline In Assessment of Growth Hormone Deficiency in Adults (AGHDA) Questionnaires at Week 36
Description: The AGHDA is a quality of life subject-administered questionnaire that is condition-specific and comprises of 25 'Yes' or 'No' statements covering 6 dimensions - mobility, pain, energy, sleep, emotional reactions and social isolation. The AGHDA total score change from Baseline values is calculated as the difference between the total score at Visit 6 (Week 36), and the total score at Baseline.
Time Frame: Baseline, Week 36
Population: Due to poor recruitment, the study was terminated early; therefore efficacy analyses were not completed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Genotropin | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in Cardiovascular Risk
Description: The cardiovascular risk parameters (low-density lipoprotein-cholesterol, high-density lipoprotein cholesterol, total cholesterol and fasting triglycerides) was measured at all visits (Weeks 2, 4, 12, 24, and 36).
Time Frame: Baseline, Weeks 2, 4, 12, 24, and 36
Population: Due to poor recruitment, the study was terminated early; therefore efficacy analyses were not completed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Genotropin | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in Weight
Time Frame: Baseline, Weeks 2, 4, 12, 24, and 36
Population: Due to poor recruitment, the study was terminated early; therefore efficacy analyses were not completed.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Genotropin | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline in Waist Circumference
Time Frame: Baseline, Weeks 2, 4, 12, 24, and 36
Population: Due to poor recruitment, the study was terminated early; therefore efficacy analyses were not completed.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Genotropin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Genotropin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 4/4 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Genotropin (N=4) | Placebo (N=6)
Pyrexia (General disorders) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.